CLINICAL TRIAL: NCT02217813
Title: A Phase 1, Open-label, Randomized, Crossover, Single Dose Study To Determine The Bioequivalence Of Pf-06291826 (Tafamidis) 20 Mg Capsule Manufactured By Catalent Versus Capsule Manufactured By Pii In Healthy Subjects Under Fasted Conditions
Brief Title: A Bioequivalence Study Comparing Two Different Tafamidis Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461044; 2014-003271-35 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Tafamidis (Experimental)
  Interventions: Drug: Tafamidis
- 2. Tafamidis (Experimental)
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 20 mg of current commercial formulation
  Other Names: Vyndaqel
  Arms: 1. Tafamidis
Drug: Tafamidis — 20 mg of new formulation
  Other Names: Vyndaqel
  Arms: 2. Tafamidis

SUMMARY:
Each subject will be given tafamidis. After swallowing a single tafamidis capsule, tafamidis blood concentrations will be measured periodically for one week. After about 20 days, subjects will take a different form of tafamidis capsule and the process repeated. Tafamidis concentrations from the two different formulations will be compared to determine if they are approximately the same.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 Kg and total body weight more than 50 Kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | 168 hours
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 168 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 168 hours
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 168 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 168 hours
Plasma Decay Half-Life (t1/2) | 168 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461044&StudyName=A%20Bioequivalence%20Study%20Comparing%20Two%20Different%20Tafamidis%20Formulations